CLINICAL TRIAL: NCT03659890
Title: The Effect of Dietary Nucleotides and Ribose on Muscle Fuel Utilisation and Exercise Performance
Brief Title: Dietary Nucleotides and Ribose on Muscle Fuel Utilisation
Acronym: FUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 171206/B/04
Record Dates: First submitted 2018-06-13; First posted 2018-09-06 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — High-Throughput Nucleotide Sequencing; Ribose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low nucleotide (Placebo Comparator): 2 week supplementation with a low nucleotide mycoprotein drink, with added dextrose
  Interventions: Dietary Supplement: Low nucleotide
- High nucleotide (Experimental): 2 week supplementation with a high nucleotide mycoprotein drink, with added dextrose
  Interventions: Dietary Supplement: High nucleotide
- High nucletide + Ribose (Experimental): 2 week supplementation with a high nucleotide mycoprotein drink, with added ribose
  Interventions: Dietary Supplement: High nucletide + Ribose

INTERVENTIONS:
Dietary Supplement: Low nucleotide — 2 week, twice daily, supplementation with a nucleotide-depleted mycoprotein drink, with added dextrose
  Arms: Low nucleotide
Dietary Supplement: High nucleotide — 2 week, twice daily, supplementation with a nucleotide-rich mycoprotein drink, with added dextrose
  Arms: High nucleotide
Dietary Supplement: High nucletide + Ribose — 2 week, twice daily, supplementation with a nucleotide-rich mycoprotein drink, with added ribose
  Arms: High nucletide + Ribose

SUMMARY:
Nucleotides are the building blocks for a variety of molecules, including ATP, which is broken down in the skeletal muscle cells to provide fuel for exercise. Nucleotides can be obtained from the diet, and produced or salvaged by the body. Though nucleotides provide the building blocks for ATP, the sugar ribose has been suggested to be rate limiting for synthesising ATP.

Previous studies have shown a decrease in ATP levels in the muscle after intense exercise, and this is linked to fatigue. Other studies have also reported benefits of nucleotide and/or ribose supplementation on exercise performance. However, any potential link between ATP metabolism and exercise performance has not been explored.

This study will look at the effects of nucleotide and nucleotide-ribose supplementation in fuel utilisation and performance in skeletal muscle during endurance exercise.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30

Exclusion Criteria:

* On medication (except contraception)
* Smokers
* Diagnosed with any metabolic or cardiovascular conditions
* Muscle or bone injuries
* BMI < 18 or > 30

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Changes in muscle ATP concentrations | After each supplementation cycle (day 15 of each cycle): baseline (fasted and before exercise), immediately after glycogen depleting exercise (after exercising for 1:30 - 2 hours), immediately after 15 minute time trial and after 3-hour recovery

SECONDARY OUTCOMES:
Changes in muscle glycogen concentrations | After each supplementation cycle (day 15 of each cycle): baseline (fasted and before exercise), immediately after glycogen depleting exercise (after exercising for 1:30 - 2 hours), immediately after 15 minute time trial and after 3-hour recovery
Blood lactate concentrations | After supplementation cycle (day 15): baseline and at 15 minute intervals up 1 hour during glycogen depleting exercise
Blood glucose concentrations | After supplementation cycle (day 15): baseline and at 15 minute intervals up 1 hour during glycogen depleting exercise
Serum uric acid concentrations | Measured at baseline and of days 6, 8 and 15 of each supplementation cycle

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter - St Luke's Campus, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No